CLINICAL TRIAL: NCT03131674
Title: The Effect of Cervical Physical Therapy Treatment in Patients With Somatic Tinnitus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Ongoing insights required a different approach
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Sarah Michiels, Post-doctoral researcher, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16/48/512
Record Dates: First submitted 2017-04-19; First posted 2017-04-27 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Tinnitus, Subjective
Keywords: Somatic tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: We use a delayed treatment design, where both groups receive the same treatment.
  One group receives the treatment immediately after the inclusion. The other group receives the treatment after a 9-weeks delay.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct treatment (Experimental)
  Interventions: Other: Cervical physical therapy
- Delayed treatment (Experimental)
  Interventions: Other: Cervical physical therapy

INTERVENTIONS:
Other: Cervical physical therapy — Patients receive a multimodal cervical physical therapy treatment

SUMMARY:
This study investigates the effect of cervical physical therapy on tinnitus annoyance in patients with somatic tinnitus. This study specifically enrolls patients with co-varying tinnitus and neck complaints, with low-pitched tinnitus or patients who's tinnitus can be influenced by neck movements or positions.

These inclusion criteria were chosen, since a prior study showed that these factors were good prognostic indicators for a positive treatment effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients with subjective tinnitus (Tinnitus Functional Index between 25 and 90 point) in combination with self-reported neck complaints (Neck Bournemouth Questionnaire > 13 points) are included in case one of the following is present:

  * Tinnitus and neck complaints increase and decrease together
  * Tinnitus is low-pitched and increases during inadequate neck postures

Exclusion Criteria:

* Tinnitus related to Ménière's disease, clear otological or neurological causes
* Serious depression
* Contra-indications for cervical spine treatment
* Patient already received cervical physical therapy in the past 2 months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Tinnitus Questionnaire | Baseline, 9 weeks, 18 weeks
  change in tinnitus distress after treatment and after follow-up

SECONDARY OUTCOMES:
Tinnitus Functional Index | Baseline, 9 weeks, 18 weeks
  change in tinnitus severity after treatment and after follow-up
Neck Bournemouth Questionnaire | Baseline, 9 weeks, 18 weeks
  change in neck complaints after treatment and after follow-up
Change in Auditory evoked potentials | Baseline, 9 weeks
  EEG measurement during auditory task
Change in Manual Rotation test | Baseline, 9 weeks
  clinical test
change in adapted Spurling test | baseline, 9 weeks
  clinical test
change in presence of active triggerpoints | baseline, 9 weeks
  clinical test
change in Craniocervical flexion test | baseline, 9 weeks
  clinical test
change in Coordination and strength test of cervical extensor muscles | baseline, 9 weeks
  clinical test
change in Speech in noise test | baseline, 9 weeks
  audiological test

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Antwerp, Edegem, Antwerp, Belgium